CLINICAL TRIAL: NCT01759641
Title: Italian Group of Study on the Role of Oxygen Saturation as a Potential Surrogate Marker of Intradialytic Cardiovascular Instability
Brief Title: Observational Study to Assess Oxygen Saturation Predictive Power Related to Intradialytic Acute Hypotension
Acronym: SOGLIA
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Antonio Santoro, Professor Antonio Santoro MD, Chief of Nephrology, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: CRC-MAL 01
Record Dates: First submitted 2012-12-24; First posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Acute Intradialytic Hypotension
Keywords: Dialysis; Monitoring; Cardiovascular stability; biosignals

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypotension-prone patients: The study group included all patients treated with standard HD prone to acute intradialytic hypotension.
  Interventions: Device: Hypotension-prone patients

INTERVENTIONS:
Device: Hypotension-prone patients — Hemox optical sensor equips the dialysis monitors used during this trial. It is able to measure continuously, on arterial blood line, oxygen saturation, hematocrit and blood volume reduction.
  Other Names: Hemox

SUMMARY:
The aim of the present work was to analyze the short-term variability of SO2 during hemodialysis in sessions with and without hypotension to correlate the SO2 variability to hemodynamic instability.

DETAILED DESCRIPTION:
During the last 40 years a lot has been achieved in dialysis regarding both monitors safety and membranes overall performances Anyway, intradialytic symptoms still remain a major concern for nephrologists: in particular, hypotension is the most frequent [1].

Intradialytic hemodynamic monitoring systems have been developed to have continuous surveillance of the main hemodynamic variables (heart rate, body temperature, blood pressure itself, cardiac output, ecc…).

In a second moment, the further evolution was towards the retroactive control systems, to force some of the variables involved in the genesis of the hemodynamic stability, along a pre-determined, ideal, trend. In this view, various bio-feedback mechanisms have been proposes along the years, for example, to tackle hypovolemia-related hypotension. Their scientific rationale is the control of either blood volume or directly natremia, in order to pilot plasma refilling towards the vascular compartment [2].

Despite the great achievements obtained, the forecasting of acute hypotension during hemodialysis still remains a complex problem, likely involving more than one variable.

SO2 can be considered an indirect expression of the hemodynamic stability. Moreover, in dialysis, it has always been regarded as a bio-compatibility marker for membranes [3]. Nowadays, SO2 changes during dialysis are easy to measure with a fully, non-invasive sensor assembled on the arterial line.

We planned this study to analyze on a large number of sessions the short-term variability of SO2 during hemodialysis in relationship with hemodynamic tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis vintage > 6 months
* Well functioning arterovenous fistula or central venous catheter
* thrice weekly HD treatment schedule
* Acute hypotensions in the last month before study start > 20% of sessions

Exclusion Criteria:

* Mental illness
* life expectancy < 6 months
* any profiling and/or biofeedback strategies routinely prescribed

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESRD patients on RRT with a recent clinical history of acute intradialytic hypotension.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
SO2 short-term variability predictive power | 3 months
  SO2 short term variability predictive power was assessed by means of common clinical tests indexes:
  sensitivity (number of sessions with effective hypotension correctly classified using SO2 standard deviation analysis)
  specificity (number of sessions without hypotension correctly classified using SO2 standard deviation analysis)

SECONDARY OUTCOMES:
Central venous catheters subgroup analysis | 3 months
  This analysis was performed, according to the method described in the Primary Outcome section, only on the group of sessions in which a central catheter was used as vascular access.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Santoro, MD, Principal Investigator — Azienda ospedaliera universitaria "S. Orsola-Malpighi", Bologna, Italy
Locations (1):
- Azienda Ospedaliero-Universitaria "S. Orsola-Malpighi", Nephrology, Dialysis and Hypertension dpt., Bologna, Italy

REFERENCES:
- [Background] Locatelli F, Altieri P, Andrulli S, Bolasco P, Sau G, Pedrini LA, Basile C, David S, Feriani M, Montagna G, Di Iorio BR, Memoli B, Cravero R, Battaglia G, Zoccali C. Hemofiltration and hemodiafiltration reduce intradialytic hypotension in ESRD. J Am Soc Nephrol. 2010 Oct;21(10):1798-807. doi: 10.1681/ASN.2010030280. Epub 2010 Sep 2. PMID 20813866
- [Background] Santoro A, Mancini E, Basile C, Amoroso L, Di Giulio S, Usberti M, Colasanti G, Verzetti G, Rocco A, Imbasciati E, Panzetta G, Bolzani R, Grandi F, Polacchini M. Blood volume controlled hemodialysis in hypotension-prone patients: a randomized, multicenter controlled trial. Kidney Int. 2002 Sep;62(3):1034-45. doi: 10.1046/j.1523-1755.2002.00511.x. PMID 12164888
- [Background] Gueler F, Gwinner W, Schiborr C, Martin M, Klos A, Kirsch T, Fiebeler A, Haller H, Fliser D. Biocompatibility parameters of different dialysis membranes assessed during systemic inflammation. Blood Purif. 2005;23(3):196-202. doi: 10.1159/000083941. Epub 2005 Feb 10. PMID 15711040